CLINICAL TRIAL: NCT05194618
Title: A Randomized, Double-blind, Parallel Groups, Placebo-controlled, Proof-of-concept Study to Assess the Efficacy and Safety of Valerian Root Extract and Lavender Essential Oil Combination in Subjects With Sleep Complaints.
Brief Title: Efficacy and Safety of Valerian Root Extract and Lavender Essential Oil Combination, Over 4 Weeks in Subjects With Sleep Complaints
Acronym: PHYTOSOM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHUBX 2021/17
Record Dates: First submitted 2021-11-30; First posted 2022-01-18 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Sleep
Keywords: Sleep; Sleep complaint; valerian; lavender

STUDY DESIGN:
Intervention Model Description: comparative, randomized, double-blind, placebo-controlled, parallel groups study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valerian/Lavender arm (Experimental): Participants in this arm will receive actives products : 420 mg per tablet of Valerian root extract and 40 mg per tablet of essential oil of Lavender
  Interventions: Dietary Supplement: Valerian - lavender
- Placebo arm (Placebo Comparator): Participants in this arm will receive placebo (no active product)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Valerian - lavender — 1 tablet per day, half hour before bedtime, day 1 to day 28
  Arms: Valerian/Lavender arm
Dietary Supplement: Placebo — 1 tablet per day, half hour before bedtime, day 1 to day 28
  Arms: Placebo arm

SUMMARY:
Several epidemiologic studies have clearly shown that sleep complaints are very common in the general population. It involves a predominant complaint of a nonrestorative sleep or dissatisfaction with sleep quality or duration and it is accompanied by difficulties in initiating sleep at bedtime, frequent or prolonged awakenings, or early-morning awakening with an inability to return to sleep.

Lavender oil as well as valerian officinalis are benefiting from a long traditional use in sleep and these products have moderate sedative effects compared to classical hypnotic compounds.

This study is proposed to assess the efficacy and the safety of this combination in subjects with slight to moderate sleep complaints.

DETAILED DESCRIPTION:
Several epidemiologic studies have clearly shown that sleep complaints are very common in the general population. It involves a predominant complaint of a nonrestorative sleep or dissatisfaction with sleep quality or duration and it is accompanied by difficulties in initiating sleep at bedtime, frequent or prolonged awakenings, or early-morning awakening with an inability to return to sleep. In a representative sample of the French population, 73% of subjects indicated the presence of a nocturnal sleep problem during the preceding month and can be considered as poor sleepers. Fifty-seven percent complained of difficulties initiating sleep 53 % complained of night awakenings, and 41 % complained of a nonrestorative sleep. Only 29% of the sample had sleep problems that would meet the diagnostic criteria for insomnia disorders defined in Diagnostic and Statistical Manual of Mental Disorders 5 (DSM5), the classification of mental disorders of the APA as difficulty to initiate or maintain sleep at least 3 times a week and for at least 3 consecutive months. Moreover, the prevalence of poor sleepers has been massively increased in the recent epidemic context.

Poor sleep is associated with increased fatigue, psychological distress, risk of suicide, higher medical costs, increased disability, and greater limitations of activity. Poor sleepers, excluding individuals with sleep-disordered breathing, other significant medical conditions and psychiatric disorders, have a potentially serious health impact. An analysis of 28 epidemiological studies found that sleep complaints are associated with psychological complaints, emotional fluctuations, alcohol and drug abuse. Health-related quality of life is nearly always affected in subjects experiencing sleep complaints (difficulty initiating or maintaining sleep), according to the findings of the large Sleep Heart Health Study.

Poor sleepers still require a medical attention. Non-medicinal methods are particularly indicated in poor sleepers: sleep hygiene advice, relaxation, restriction of time spent in bed, and cognitive-behavioural therapies that combine these approaches. In poor sleepers, use complementary health approaches such as herbal to promote or maintain sleep must also receive the most research attention.

As single ingredients, valerian officinalis root extract has been identified as having clinical evidence to demonstrate improvement in insomnia complaints:

* Sleep onset latency
* Night awakenings
* Sleep quality
* Sleep efficiency Studies have also demonstrated that Lavandula angustifolia essential oil had a beneficial effect on anxiety and disturbed sleep.

Lavender oil as well as valerian officinalis are benefiting from a long traditional use in sleep and these products have moderate sedative effects compared to classical hypnotic compounds.

The existing published clinical trials as well as the traditional use suggest a positive effect on sleep and stress, however Valerian aqueous extract and lavender essential oil have been studied in the past for different dosages, for small simple size and standalone only.

Therefore it is difficult to fully rely on the past literature to estimate the potential effect of the combination Valerian - Lavender Essential Oil, that explain the purpose of this proof of concept study which aim to better quantify the effect of the combination on sleep complaints compared to a placebo group in the targeted population.

This study is proposed to assess the efficacy and the safety of this combination in subjects with slight to moderate sleep complaints.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (≥ 18 years old) with sleep complaints:

   * with a frequency of 1 or 2 times per week, OR
   * with a frequency ≥ 3 times per week and duration < 3 months,

   Sleep complaints are defined as:
   * Difficulty initiating sleep, or
   * Difficulty maintaining sleep, or
   * Early-morning awakening with inability to return to sleep. and
   * Causing distress or impairment in social, occupational, educational, academic, behavioral, or other important areas of functioning.
2. Insomnia Severity Index (ISI) score comprised between 11 and 21 (slight to moderate sleep complaints)
3. BMI inferior to 30 (included)
4. Connected to internet and having a smartphone
5. Affiliated person or beneficiary of a social security scheme
6. Free, informed and written consent signed

Exclusion Criteria:

1. Severe sleep complaints (ISI > 21) OR insomnia with clinical significance consequences as defined by DSM 5
2. Subject with other organic sleep disorders diagnosed (i.e. sleep apnea, Restless Legs Syndrome)
3. Subject at high risk of suspicion of Obstructive Sleep Apnea Syndrome (OSAS) on the STOP-BANG questionnaire (Snoring, Tiredness, Observed apnea, blood Pressure, Body mass index, Age, Neck circumference and Gender), or a suspicion of Restless Legs Syndrome (RLS) on the RLS screening questionnaire,
4. Subject with a significant medical history in the previous year or still in progress (example: Cancer),
5. Subject with acute psychiatric disorder (mood disorders, severe anxiety disorders, psychosis, addiction interfering with nocturnal sleep). Subject with a history of mood or anxiety disorder currently stabilized could be included.
6. Having initiated a psychotropic treatment for anxiety or mood disorders in the last 2 months or whose treatment dose has been modified for less than 2 months (antidepressant, anxiolytic and antihistamine treatments will be allowed if they are prescribed for a stabilized mood and/or anxiety disorder)
7. Having organic disorders inducing sleep complaints (i.e. Covid < 6 months)
8. Currently treated for insomnia disorders with a pharmaceutical treatment (hypnotic treatments, anxiolytic, antidepressants).
9. Taking food supplements aimed at improving sleep quality in the previous month,
10. Taking food supplements in the previous month containing valerian root extract or lavender oil
11. Taking any pharmaceutical treatment suspected to induce sleep complaints
12. Shift workers and social jet lag
13. Having undertaken trans-meridian travel (± 3H) in the previous month and/or refusing not to undertake trans-meridian travel (± 3H) )
14. Known drug abuse
15. Alcohol consumption more than 10 standard drinks per week
16. Caffeine consumption more than 5 standard cups/drinks per day
17. Participation in a clinical trial in the previous 3 months that may interfere with the evaluation of the primary endpoint (sleep complaints) or exclusion period still on going
18. Eating disorders: anorexia and bulimia or unstable dietary pattern;
19. Any food allergy documented or suspected to one of the components of the study products;
20. Pregnancy or breast-feeding woman (contraceptive mandatory)
21. Subject under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | Day28 after inclusion (Day1)
  The Insomnia Severity Index is a 7-item self-administered questionnaire asking about difficulties sleeping and thoughts and worries about sleep.
  A 5-point scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28.
  The total score is interpreted as follows:
  * absence of insomnia (0-7);
  * sub-threshold insomnia (8-14);
  * moderate insomnia (15-21); and
  * severe insomnia (22-28).

SECONDARY OUTCOMES:
Sleep onset latency | Change from baseline (Day 1) to end of supplementation (Day 28)
  Duration of time in minutes from turning the light off to falling asleep
Sleep efficiency | Change from baseline (Day 1) to end of supplementation (Day 28)
  ratio of total sleep time to time in bed
Wake after sleep onset | Change from baseline (Day 1) to end of supplementation (Day 28)
  Wake after sleep onset in minutes
Total sleep time | Change from baseline (Day 1) to end of supplementation (Day 28)
  Total sleep time in minutes
Time in bed | Change from baseline (Day 1) to end of supplementation (Day 28)
  Time in bed in minutes
Perceived quality of sleep using Leeds Sleep Evaluation Questionnaire (LSEQ) | end of supplementation (Day 28)
  The Leeds Sleep Evaluation Questionnaire (LSEQ)(48) assesses 4 consecutive aspects of sleep: getting to sleep, quality of sleep, awakening from sleep, and behaviour following wakefulness.
  It is self-administered and contains 10 items related to the 4 aspects of sleep. The participant is asked to answer the questions by placing a mark vertically on a 100mm length visual analogue scale. The score for each of the 4 aspects of sleep is the mean of the ratings for each aspect.
  The questionnaire is used to monitor subjectively perceived changes in sleep during psychopharmacological interventions.
Change from baseline to 4 weeks in Hospital Anxiety and Depression Scale (HADS) scores | Change from baseline (Day 1) to end of supplementation (Day 28)
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item self-report measure of anxiety and depression symptoms. The HADS comprises 14 items each rated from 0 to 3, with higher scores indicating greater anxiety/depression. The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states. The anxiety and depression subscales each have seven items and a maximum score of 21.
SF-36 mental and physical scores | Change from baseline (Day 1) to end of supplementation (Day 28)
  The Short-Form Health Survey (SF-36) is a 36-item general health-related quality of life measure. It measures 8 general health concepts: physical functioning, role physical, bodily pain, general health, vitality, social functioning role emotional and mental health. These concepts are summarized as physical and mental components scores.
  Higher scores indicate better health status.
FOSQ-10 scores | Change from baseline (Day 1) to end of supplementation (Day 28)
  The Functional Outcomes of Sleep Questionnaire (FOSQ), has been used in research and clinical practice to measure the impact of daytime sleepiness on activities of daily living. This questionnaire includes 30 items.
  A shorter version of the instrument, including only 10 items (FOSQ-10) that may be more easily implemented in clinical practice, has been developed. These 10 questions are distributed among 5 subscales as follows: general productivity (2 item), activity level (3 items), vigilance (3 items), social outcomes (1 item) and sexual relationship (1 item). Items have to be rated on a scale of 1-4 (1 = extreme difficulty, 2 = moderate difficulty, 3 = a little difficulty, 4 = no difficulty).
  The total score is the sum of the 5 sub scores.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No